CLINICAL TRIAL: NCT05661539
Title: The Effect of Baseline and First Trimester Uterine Artery Doppler Velocimetry Parameters on Obstetric Outcomes in HRT-FET Cycles: Prospective Cohort Study
Brief Title: Baseline and First Trimester Uterine Artery Doppler Velocimetry to Predict Poor Obstetric Outcomes in IVF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, ŞAFAK OLGAN, Associate Professor, Akdeniz University
Other Study IDs: 49829698
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Infertility, Female
Keywords: Uterine Artery Doppler Velocimetry; Baseline Uterine Artery Doppler Velocimetry; First Trimester Uterine Artery Doppler Velocimetry
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- non-pregnant: negative b-hCG results 9 days after embryo transfer.
  Interventions: Device: Transvaginal Ultrasonography
- pregnant with obstetric complications: Patients with a positive pregnancy result who develop obstetric complications such as preeclampsia, eclampsia, fetal growth restriction, oligohydramnios, polyhydramnios, preterm birth, gestational diabetes mellitus, antenatal bleeding and etc. after the 20th gestational weeks.
  Interventions: Device: Transvaginal Ultrasonography
- pregnant without obstetric complications: Patients who have positive pregnancy results and do not have any obstetric complications such as preeclampsia, eclampsia, fetal growth restriction, oligohydramnios, polyhydramnios, preterm birth, gestational diabetes mellitus, antenatal bleeding and etc. during pregnancy.
  Interventions: Device: Transvaginal Ultrasonography

INTERVENTIONS:
Device: Transvaginal Ultrasonography — The amount of resistance and blood flow in the main arteries that provide uterine perfusion will be determined by uterine artery Doppler velocimetry performed on the patients.

SUMMARY:
The researchers aim to determine how baseline (preconceptional) and first-trimester uterine artery Doppler measurements affect obstetric complications in women undergoing high-quality blastocyst transfer and to determine the correlation between the two Doppler measurements.

DETAILED DESCRIPTION:
Only patients with high-quality blastocyst-stage embryos will be included in the study. In frozen embryo transfer cycles prepared hormonally, basal bilateral uterine artery Doppler velocimetry will be performed before treatment (preconception) in each patient.

Bilateral uterine artery Doppler velocimetry will be performed during the basal ultrasonography (2-5 days of menstruation). The absence of any uterine artery notches, diastolic or reverse flow will also be noted. In addition, sub-endometrial (arcuate artery) blood flows will be evaluated by Doppler ultrasonography.

For endometrial preparation, estrogen replacement will be given for approximately 12-14 days as a routine In cases with endometrial thickness ≥7mm, progesterone treatment will be started and embryo transfer will be planned on the 6th day of the treatment.

In the pregnant group, measurements will be repeated at the end of the first trimester (11-14 weeks) and uterine artery Doppler velocimetry will be reevaluated. In addition, patients will be followed up until delivery and possible obstetric complications will be recorded.

Baseline and first-trimester uterine artery Doppler ultrasonography findings will be compared with obstetric results. Obstetric outcomes such as birth weight at the end of pregnancy, small-large for gestational age, presence of hypertension, and preterm delivery will be correlated with preconceptional and first-trimester uterine artery Doppler parameters.

ELIGIBILITY:
Inclusion Criteria:

* Exogenous hormone preparation of the endometrial lining
* High embryo quality ((≥2BB) according to Alpha criteria
* Embryo transfer at the blastocyst stage

Exclusion Criteria:

* Patients whose treatments were canceled for any reason before the embryo transfer procedure
* Patients who underwent embryo transfer in the cleavage stage
* Presence of low-quality (<2BB) blastocysts
* >15% loss of viability of the embryo during embryo thawing,
* Patients with congenital uterine malformations,
* Patients in whom Doppler velocimetry cannot be performed optimally

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: All patients who have artificial endometrial preparation with high-quality blastocysts between May 2022 and December 2022 will be included.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Live Birth Rate | 9 months
  pregnancy beyond 24 weeks of gestational age.
Obstetric Complication Rates | 20 weeks after embryo transfer
  Conditions such as preeclampsia, eclampsia, fetal growth restriction, oligohydramnios, polyhydramnios, preterm birth, gestational diabetes mellitus, antenatal bleeding and etc. that develop during pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: ŞAFAK OLGAN, MD, Principal Investigator — Akdeniz University; ARİF ÖZSİPAHİ, MD, Study Chair — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)